CLINICAL TRIAL: NCT03390647
Title: A Phase 1 Clinical Study of E6130 - Clinical Pharmacology Study in Healthy Adult Male Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics in Healthy Adult Male Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision of Sponsor
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: E6130-CP2
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Healthy Participants
Keywords: E6130; Healthy adult male participants; Phase 1; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A1 (Experimental): Japanese participants will receive a single oral dose of E6130 on Day 1 and Day 7 administered in the specified order (fasted/fed or fed/fasted) to evaluate the food effect.
  Interventions: Drug: E6130
- Cohort B1 (Experimental): Caucasian participants will receive a single oral dose of either E6130 or placebo on Day 1.
  Interventions: Drug: E6130; Drug: Placebo
- Cohorts A2-A4 (Experimental): Japanese participants will receive multiple oral doses of E6130 or placebo on Days 1 to 5, administered in a randomized, dose-ascending manner.
  Interventions: Drug: E6130; Drug: Placebo

INTERVENTIONS:
Drug: E6130 — Oral dose
Drug: Placebo — E6130-matched placebo
  Arms: Cohort B1; Cohorts A2-A4

SUMMARY:
The primary purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of multiple oral doses of E6130 in Japanese healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in this study.

1. Japanese or Caucasian healthy adult males aged ≥20 and <45 years at the time of informed consent who are non-smokers or able to stop smoking from at least 4 weeks before study drug administration until the post-treatment examination
2. Has voluntarily consented, in writing, to participate in this study
3. Has been thoroughly briefed on the conditions for participation in the study, and are willing and able to comply with the conditions

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study.

1. History of surgical treatment may affect the pharmacokinetics of the study drug at screening
2. Suspected to have clinically abnormal symptoms or impairment of organ function requiring treatment on the basis of history and complications at screening, and physical findings, vital signs, electrocardiogram findings, or laboratory values at screening or baseline
3. History of drug allergy at screening
4. Judged by the investigator or sub investigator to be inappropriate for participation in this study

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) as a measure of safety and tolerability | Days 1 to 14 (Cohort A1); Days 1 to 12 (Cohorts A2 to A4); Days 1 to 8 (Cohort B1)

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of E6130 | Days 1 to 4 and Days 7 to 10 (Cohort A1); Days 1 to 4 (Cohort B1)
Maximum observed serum concentration at steady state (Css, max) of E6130 | Days 1 to 7 (Cohorts A2 to A4)
Time to Cmax (tmax) of E6130 | Days 1 to 4 and Days 7 to 10 (Cohort A1); Days 1 to 4 (Cohort B1)
Time to Cmax at steady state (tss, max) of E6130 | Days 1 to 7 (Cohorts A2 to A4)
Area under the serum concentration-time curve from zero time to the time of last quantifiable concentration (AUC[0-t]) of E6130 | Days 1 to 4 and Days 7 to 10 (Cohort A1); Days 1 to 4 (Cohort B1)
Area under the serum concentration-time curve from zero time extrapolated to infinite time (AUC[0-inf]) of E6130 | Days 1 to 4 and Days 7 to 10 (Cohort A1); Days 1 to 4 (Cohort B1)
Area under the serum concentration-time curve from zero time to 24 hours (AUC[0-24h]) of E6130 | Days 1 to 7 (Cohorts A2 to A4)
Terminal elimination phase half-life (t1/2) of E6130 | Days 1 to 7 (Cohorts A2 to A4)